CLINICAL TRIAL: NCT04364425
Title: Comparing Low Dose and High Dose Steroid Injection for Adhesive Capsulitis
Brief Title: Steroid Injection for Adhesive Capsulitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-07-005C
Record Dates: First submitted 2020-04-20; First posted 2020-04-28 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Adhesive Capsulitis
MeSH Terms: conditions — Bursitis | interventions — Triamcinolone Acetonide; Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low dose steroid (Experimental): patient received ultrasound-guided 40mg triamcinolone + 4cc xylocaine + 12cc NS
  Interventions: Drug: Triamcinolone Acetonide; Drug: lidocaine hydrochloride; Drug: Normal saline
- high dose steroid (Active Comparator): patient received ultrasound-guided 10mg triamcinolone + 4cc xylocaine + 15cc NS
  Interventions: Drug: Triamcinolone Acetonide; Drug: lidocaine hydrochloride; Drug: Normal saline

INTERVENTIONS:
Drug: Triamcinolone Acetonide — ultrasound guided steroid injection using 1ml of 10mg or 4ml of 40mg triamcinolone acetonide
  Other Names: triamcinolone acetonide 10mg/ml (Shincort, YSP, Taiwan)
Drug: lidocaine hydrochloride — Ultrasound guided injection using 4ml of 2% lidocaine hydrochloride (Xylocaine)
  Other Names: lidocaine hydrochloride (Xylocaine)
Drug: Normal saline — Ultrasound guided injection using 15ml or 12 ml of normal saline

SUMMARY:
This study was conducted to compare the efficacy of hydrodilatation with low dose steroid with high dose steroid for treating adhesive capsulitis.

DETAILED DESCRIPTION:
Design: a prospective, double-blinded, randomized, clinical trial

Patient and methods:

Patients with adhesive capsulitis for at least 3 months were enrolled and randomly allocated into group 1 (hydrodilatation with low dose steroid ) and group 2 (hydrodilatation with high dose steroid). The patients were evaluated before treatment and were reevaluated 0, 6, and 12 weeks after the beginning of the treatment. Outcomes measures included a pain scale (visual analog scale), range of motion, Constant shoulder score, Shoulder Pain And Disability Index

ELIGIBILITY:
Inclusion Criteria:

1. clinical diagnosis of adhesive capsulitis
2. a duration of complaints more than 3 months
3. a reduction in passive range of motion in at least 2 of the following: forward flexion, abduction, or external rotation of the affected shoulder of more than 30 degree compared with the other side.

Exclusion Criteria:

1. prior manipulation of the affected shoulder under anesthesia;
2. other conditions involving the shoulder ( rheumatoid arthritis, Hill-Sachs lesions, osteoarthritis, damage to the glenohumeral cartilage,osteoporosis, or malignancies in the shoulder region);
3. neurologic deficits affecting shoulder function in normal daily activities;
4. shoulder pain caused by cervical radiculopathy
5. a history of drug allergy to hyaluronic acid;
6. pregnancy or lactation;
7. received injection into the affected shoulder during the preceding 3 months

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-05-04 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
change in pain intensity | 0, 6, 12 wks.
  pain intensity was measured by visual analog scale (0-10)

SECONDARY OUTCOMES:
change in Shoulder Pain And disability index | 0, 6, 12 wks.
  The Shoulder Pain and Disability Index (SPADI) is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities. The pain dimension consists of five questions regarding the severity of an individual's pain. Functional activities are assessed with eight questions designed to measure the degree of difficulty an individual has with various activities of daily living that require upper-extremity use. The SPADI takes 5 to 10 minutes for a patient to complete and is the only reliable and valid region-specific measure for the shoulder.
change in glenohumeral joint range of motion | 0, 6, 12 wks.
  Shoulder flexion, abduction, external rotation and internal rotation were measured with goniometer with patient in supine position.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei veteran general hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Wang JC, Hsu PC, Wang KA, Wu WT, Chang KV. Comparative Effectiveness of Corticosteroid Dosages for Ultrasound-Guided Glenohumeral Joint Hydrodilatation in Adhesive Capsulitis: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2023 May;104(5):745-752. doi: 10.1016/j.apmr.2022.11.007. Epub 2022 Dec 12. PMID 36521580